CLINICAL TRIAL: NCT04502160
Title: The Northern Ireland Haemodialysis Vascular Access Database
Acronym: NIVAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19089JH-SS
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Hemodialysis Access Failure; Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vascular Access Creation — arteriovenous fistula creation
  Other Names: arteriovenous fistula creation

SUMMARY:
This is database designed to explore clinical outcomes related to vascular assess in the population of Northern Ireland with CKD Stage 5 and End-stage Renal Failure.

DETAILED DESCRIPTION:
Vascular access is the conduit by which blood is transferred from the patient to the dialysis machine and back to the patient during therapy. There are three types of vascular access: Arteriovenous fistulas (AVF), Central venous catheters (CVC) and Arteriovenous grafts (AVG).

AVFs are associated with the best patient survival in individuals undergoing dialysis therapy. However, Up 30-50% of AVFs thrombose or fail to mature sufficiently to support dialysis.

The aim of this database is to further research in the area of AVF outcomes using routinely collected clinical data..

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending Nephrology undergoing AVFcreation between January 2009 and December 2019 in a single centre (Belfast City Hospital

Exclusion Criteria:

* None

Ages: 16 Years to 105 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals undergoing AVF creation between January 2009 and December 2020 in a single centre (Belfast City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-10-22 (Estimated); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Rates of Arteriovenous Fistula Failure to Mature | 1 year
  Rates of Arteriovenous Fistula Failure to Mature

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hanko, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast City Hospital, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Would require application to Belfast Health and Social Care Trust Research and Development office